CLINICAL TRIAL: NCT04600167
Title: A Randomized Double Blind Placebo Controlled Trial of Rifapentine and Isoniazid for Prevention of Tuberculosis in People With Diabetes
Brief Title: Preventive Treatment Of Latent Tuberculosis Infection In People With Diabetes Mellitus
Acronym: PROTID
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Nyanda Elias Ntinginya (Other Government)
Collaborators: Stichting Katholieke Universiteit- Radboudumc (RUMC), Netherlands (Unknown); Otago University, New Zealand (Unknown); Makerere University (Other); St George's, University of London, United Kingdom (Unknown); Kilimanjaro Christian Medical University College (KCMUCo), Tanzania (Unknown); Uganda Martyrs Hospital Lubaga, Uganda (Unknown); King's College London (Other)
Responsible Party: Sponsor-Investigator, Dr. Nyanda Elias Ntinginya, Director, NIMR - Mbeya Medical Research Centre, National Institute for Medical Research, Tanzania
Organization: National Institute for Medical Research, Tanzania (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIMR-MB-002
Record Dates: First submitted 2020-09-15; First posted 2020-10-23 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus; Tuberculosis
Keywords: Tuberculosis; Drugs; Social science; Health systems; Epidemiology; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Tuberculosis | interventions — Isoniazid; rifapentine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isoniazid and Rifapentine (INH-RPT) (Experimental): Participants in intervention arm will receive an oral combination of rifapentine (RPT, 900 mg) and isoniazid (INH, 900 mg), once-weekly for 12 weeks.
  Interventions: Drug: Isoniazid and Rifapentine (INH-RPT)
- Control (Placebo Comparator): Participants in the control arm will receive placebo once weekly for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isoniazid and Rifapentine (INH-RPT) — Oral combination of rifapentine (RPT, 900 mg) and isoniazid (INH, 900 mg), once-weekly for 12 weeks.
  Other Names: 3HP
  Arms: Isoniazid and Rifapentine (INH-RPT)
Drug: Placebo — Participants in the control group will receive placebo once weekly for 12 weeks
  Arms: Control

SUMMARY:
Diabetes mellitus (DM) increases susceptibility to Tuberculosis (TB) and worsens TB patient outcomes. The number of patients with combined TB and DM now outnumbers that of combined TB and HIV and it has been estimated that 15-30% of TB disease may be attributable to diabetes globally. This may be expected to rise substantially as DM prevalence increases. Treatment of Latent TB Infection (LTBI) in this population will likely have a significant clinical benefit. Similar to HIV-infected individuals, those with DM might benefit from therapy to prevent the development of TB disease. Current international guidelines do not recommend LTBI management in people with DM, but this is because no studies have examined the risk-benefit ratio of such an intervention. To date, no RCTs have been conducted to investigate the efficacy and safety of preventive treatment of LTBI in DM patients. Based on evidence on effectiveness, safety, and treatment completion rates, 3HP has been selected as the regimen of choice for this study of African people living with DM. People living with DM will be randomized to 3HP or placebo to determine the efficacy of 3HP in the prevention of TB disease in this population. PROTID's preventive treatment of LTBI among people with DM will generate the first solid evidence to support or refute the use of preventive treatment against TB in people with DM.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in diabetes care with a history of DM and current use of anti-diabetic medication ('known DM'); OR in the absence of anti-diabetic medication an HbA1c of =6.5% (48 mmol/mol) or a fasting venous plasma glucose of =7.0 mmol (126 mg/dl). For those with no previously known DM a repeat test above the diagnostic cut-point is required to confirm the diagnosis ('new DM')
2. Adult (18 years or older)
3. Diagnosed with LTBI, defined as a positive IGRA test or TST reactivity =10 mm
4. Voluntarily signed Informed Consent Form
5. If sexually active, willing to use an effective contraceptive method for the duration of preventive therapy.

Exclusion Criteria:

1. Weight <45 kg
2. Previous TB disease, defined as either bacteriologically confirmed or clinically diagnosed and treated
3. Treatment with a rifamycin medication or isoniazid in the previous 2 years.
4. Diagnosis of probable or definite TB during screening
5. Confirmed HIV-infection or receiving antiretroviral treatment
6. Liver dysfunction, defined as serum aspartate aminotransferase (AST) level 5 times the upper limit of normal
7. Pregnant or planning to become pregnant in the next 3 months, or lactating
8. Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation
9. Other conditions inapplicable for participation in this study, such as likely to fail to adhere to study commitment or to complete the whole study, at the discretion of the site investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
First diagnosis of TB | Through study completion, median of 33 months follow-up
  The primary outcome will compare the rate of occurrence of TB disease (defined as definite or probable TB) in treatment and control groups. Definite TB disease will be confirmed by a culture or Xpert positive result for M. tuberculosis. Probable TB will be diagnosed according to an algorithm that takes into account symptoms, chest x-ray reading, sputum smear, histology and verbal autopsy results.

SECONDARY OUTCOMES:
Occurrence of possible, probable or definite TB disease | At least 24 months post randomisation
Occurrence of an adverse event | From randomisation to 60 days after end of study treatment
Treatment completion | Defined as > 11 of 12 doses of treatment over no more than 16 weeks.
All-cause mortality | At least 24 months post randomisation
Occurrence of possible, probable, or definite TB, or death | At least 24 months post randomisation
  Occurrence of possible, probable, or definite TB, or death, noting that a proportion of deaths are likely to be due to TB but not possible to confirm through verbal autopsy and clinical notes review.

CONTACTS AND LOCATIONS:
Overall Officials: Nyanda E Ntinginya, MD, MSc., Ph.D, Study Chair — Mbeya Medical Research Center, National Institute for Medical Research, Tanzania; Nyasatu Chamba, MD., Principal Investigator — Kilimanjaro Christian Medical Centre,Moshi,Tanzania; Irene Andia- Biraro, MD., Ph.D., Principal Investigator — Makerere University, Makerere, Uganda; Davis Kibirige, MD, Ph.D., Principal Investigator — Martyrs Hospital Lubaga, Makerere, Uganda
Locations (4):
- Tanzania (2):
  - Mbeya zonal referral hospital, Mbeya
  - Kilimanjaro Christian Medical Center, Moshi
- Uganda (2):
  - Makerere University, Kampala
  - Martyrs Hospital Lubaga, Kampala

REFERENCES:
- [Derived] Ntinginya NE, Te Brake L, Sabi I, Chamba N, Kilonzo K, Laizer S, Andia-Biraro I, Kibirige D, Kyazze AP, Ninsiima S, Critchley JA, Romeo R, van de Maat J, Olomi W, Mrema L, Magombola D, Mwayula IH, Sharples K, Hill PC, van Crevel R; PROTID Consortium. Rifapentine and isoniazid for prevention of tuberculosis in people with diabetes (PROTID): protocol for a randomised controlled trial. Trials. 2022 Jun 10;23(1):480. doi: 10.1186/s13063-022-06296-8. PMID 35689272
- [Derived] Olomi W, Andia Biraro I, Kilonzo K, Te Brake L, Kibirige D, Chamba N, Elias Ntinginya N, Sabi I, Critchley J, Sharples K, Hill PC, Van Crevel R. Tuberculosis Preventive Therapy for People With Diabetes Mellitus. Clin Infect Dis. 2022 Apr 28;74(8):1506-1507. doi: 10.1093/cid/ciab755. No abstract available. PMID 34505132